CLINICAL TRIAL: NCT05555355
Title: A Prospective, Single-center Study for the Investigation of the Use of Prevena Vacuum-Assisted Closure Devices in Patients Undergoing Spine Surgery
Brief Title: Prevena Spine for Use in Spine Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: 3M (Industry)
Responsible Party: Principal Investigator, Robert Galiano, Associate Professor of Surgery, Northwestern University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00216293
Record Dates: First submitted 2022-05-04; First posted 2022-09-26 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Surgery; Incision, Surgical
Keywords: negative pressure wound therapy; incisional wound therapy; spine surgery
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Intervention Model Description: Single center study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1 (control) (Placebo Comparator): Prospective control of patients who did not use Prevena following spine surgery.
  Interventions: Procedure: Spine surgery
- Group 2 (Prevena) (Active Comparator): Prospective group of patients receiving spine surgery who will have Prevena applied to incision area.
  Interventions: Device: Prevena Plus 125 Therapy Unit; Procedure: Spine surgery

INTERVENTIONS:
Device: Prevena Plus 125 Therapy Unit — The investigators will utilize the KCI USA, Inc Prevena Plus 125 vacuum-assisted closure device in patients undergoing spine surgery as a method to prevent surgical site infections and wound dehiscence after surgery. The device has been approved by the FDA under the name "Prevena 125 and Prevena Plus 125 Therapy Units" and regulation number 21CFR 878.4783.
  Arms: Group 2 (Prevena)
Procedure: Spine surgery — Patients will receive spine surgery

SUMMARY:
A pilot, prospective, single-center study for the investigation of the use of Prevena Vacuum-Assisted Closure devices in patients undergoing spine surgery.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the efficacy of the Prevena Plus 125 therapy Unit (KCI USA, Inc.) in preventing surgical site infections and other wound complications in patients undergoing spine surgery compared to conventional wound dressing. Furthermore, the investigators want to illustrate which patients benefit most significantly from Prevena usage as spine surgery sees a range of potential candidates, and not all may experience equivalent recovery from spine surgery with Prevena intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing spinal fusion surgery
2. Over 18 years old

Exclusion Criteria:

1. Medical or psychiatric condition that may increase the risk with study participation, may complicate patient compliance, or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study
2. Subjects who are pregnant at the date of surgery (SOC for surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Frequency of Surgical site infections | 1-6 weeks following surgery
  Determine if infection is present at surgical site or not.
Frequency of Wound dehiscence | 1-6 weeks following surgery
  Determine if wound reopening (dehiscence) is present at surgical site or not.
Frequency of Seroma | 1-6 weeks following surgery
  Determine if seromas (collection of fluid under the skin) are present at surgical site or not.

SECONDARY OUTCOMES:
Frequency of skin necrosis | 1-6 weeks following surgery
  Measure the frequency of patients who experience skin necrosis in the incision area
Frequency of readmission | 1-6 weeks following surgery
  Measure the frequency of patients who are readmitted following surgery due to wound-related complications

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No